CLINICAL TRIAL: NCT07403461
Title: Comparative Effects of High-Intensity Interval Training Modalities on Physical Performance and Physiological Responses in Competitive Table Tennis Players
Brief Title: HIIT Effects on Table Tennis Players
Acronym: HIIT-TTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Alirıza Han Civan, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: / E-77192459-050.99-376986
Record Dates: First submitted 2026-01-16; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Physical Fitness; Neuromuscular Function; Exercise Performance
Keywords: High-Intensity Interval Training (HIIT); Tabata Training; Physiological Adaptations; Neuromuscular Performance; Table Tennis Athletes

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to receive different Tabata-based high-intensity interval training (HIIT) modalities alongside their regular table tennis training. Assessments were conducted pre- and post-intervention to evaluate neuromuscular and physiological adaptations.
Masking Description: No masking was implemented; participants, trainers, and assessors were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calisthenic/Plyometric HIIT Group (Experimental): Participants in this group perform a Tabata-based high-intensity interval training program focused on calisthenic and plyometric exercises, in addition to their regular table tennis training. Sessions are conducted three times per week for eight weeks.
  Interventions: Behavioral: Calisthenic/Plyometric HIIT; Behavioral: Kettlebell HIIT
- Kettlebell HIIT Group (Experimental): Participants in this group perform a Tabata-based high-intensity interval training program focused on kettlebell exercises, in addition to their regular table tennis training. Sessions are conducted three times per week for eight weeks.
  Interventions: Behavioral: Calisthenic/Plyometric HIIT; Behavioral: Kettlebell HIIT

INTERVENTIONS:
Behavioral: Calisthenic/Plyometric HIIT — Participants perform a high-intensity Tabata protocol focusing on calisthenic and plyometric exercises designed to improve agility, flexibility, vertical jump performance, and neuromuscular function. Each session lasts 20-30 minutes, three times per week for eight weeks, in addition to regular table tennis training.
  Other Names: Tabata-style Calisthenic HIIT
Behavioral: Kettlebell HIIT — Participants perform a high-intensity Tabata protocol focusing on kettlebell exercises designed to improve sprint performance, VO₂max, and overall physiological adaptations. Each session lasts 20-30 minutes, three times per week for eight weeks, in addition to regular table tennis training.
  Other Names: Tabata-style Kettlebell HIIT

SUMMARY:
This study aims to investigate the effects of two different Tabata-based high-intensity interval training (HIIT) modalities on neuromuscular and physiological performance in competitive table tennis players. Participants will be randomly assigned to either a calisthenic/plyometric HIIT group or a kettlebell-based HIIT group. Both groups will perform their respective training protocols in addition to regular table tennis training for eight weeks. Physical performance and physiological variables will be assessed before and after the intervention.

DETAILED DESCRIPTION:
This study is designed as a randomized parallel-group interventional trial to examine the effects of two different Tabata-based high-intensity interval training (HIIT) modalities on neuromuscular and physiological parameters in competitive table tennis players.

Twenty-four male athletes aged between 18 and 24 years will be randomly assigned to one of two groups: a calisthenic/plyometric HIIT group or a kettlebell-based HIIT group. Both groups will continue their regular table tennis training and additionally perform their assigned HIIT protocol three times per week for a total duration of eight weeks.

The calisthenic/plyometric HIIT program consists of bodyweight and plyometric exercises performed in a Tabata format, while the kettlebell HIIT program consists of resistance-based exercises using kettlebells performed in the same interval structure. Each training session lasts approximately 20-30 minutes.

Outcome measures will be assessed before and after the intervention period and will include agility, flexibility, vertical jump performance, sprint performance, peak and average power output, and maximal oxygen uptake (VO₂max).

ELIGIBILITY:
Inclusion Criteria:

* Male table tennis athletes aged 18-24 years.
* Minimum of 2 years of regular competitive table tennis experience.
* Currently performing structured training at least 3 days per week.
* Medically cleared for high-intensity exercise.
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Any chronic illness or cardiovascular/metabolic disorders.
* Musculoskeletal injury within the last 6 months that limits physical activity.
* Participation in other high-intensity training programs outside the study protocol during the intervention.
* Inability to complete at least 90% of the scheduled intervention sessions.
* Signs of acute injury, excessive fatigue, or cardiovascular abnormalities during screening.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-11-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-03 (Actual)

PRIMARY OUTCOMES:
Agility Performance (seconds) | Pre-intervention and post-intervention (8 weeks)
  Agility will be assessed using a standardized T-test protocol to measure change-of-direction speed.
Flexibility (cm) | Pre-intervention and post-intervention (8 weeks)
  A sitting and reaching test will be used to assess lower body flexibility.

SECONDARY OUTCOMES:
Vertical Jump Height (cm) | Pre-intervention and post-intervention (8 weeks)
  Vertical jump performance will be measured using a countermovement jump test performed on a jump mat.
Sprint Performance - 10 m (seconds) | Pre-intervention and post-intervention (8 weeks)
  Sprint performance will be assessed over a distance of 10 meters using electronic timing gates.
Peak Power Output (Watts) | Pre-intervention and post-intervention (8 weeks)
  Peak power output will be measured using a standardized lower-body power assessment.
Maximal Oxygen Uptake (VO₂max) (ml/kg/min) | Pre-intervention and post-intervention (8 weeks)
  Maximal oxygen uptake (VO₂max) will be assessed using a graded exercise test performed on a treadmill or cycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Alirıza Han Civan, Dr, Study Director — Karabük Üniversitesi Hasan Doğan Spor Bilimleri Fakültesi Spor Yöneticiliği Bölümü
Locations (1):
- Karabük University, Karabük, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2026-01-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT07403461/Prot_000.pdf